## Official Title of the study:

## A Randomized Controlled Trial with Rituximab for Psychotic Disorder in Adults (RCT-RITS)

## NCT05622201

The 3.1 version of the study protocol was approved by the Ethical committee, Stockholm, Sweden on the 30<sup>th</sup> of August 2023 and by the Swedish medical product agency on the 8<sup>th</sup> of August 2023.

## Consent to participate in the study

I have received oral and written information about the study and have had the opportunity to ask questions. I get to keep the written information.

| | | | Yes | No |
|---|---|---|---|---|
| | <ul> <li>I agree to participate in the study RCT-RITS, Rituximab – a placebo-controlled study for psychosis</li> </ul> | | | |
| N | Meaning: | | | |
| | a. I consent to data about me being processed in the manner described in the research subject information. | | | |
| | <ul> <li>b. I agree that the study monitor have access to medical<br/>records for checking the data.</li> </ul> | | | |
| С | c. I agree that the research group have access to my data. | | | |
| | | | Yes | No |
| | I agree to provide samples of spinal fluid through lumbar puncture and that these are saved in the biobank. | | | |
| | <ul> <li>I agree to blood samples being taken and stored in a biobank in the<br/>manner described in the research subject information.</li> </ul> | | | |
| | I agree to undergo MRI examination in the manner described in the research subject information. | | | |
| | I agree that relatives or other persons who know me well can be interviewed about my state of health and fill out a questionnaire | | | |
| aft | er I receive the treatment. | | | |
| • la | I agree to be interviewed about my experiences of the study | | | |
| after treatment and answer a short questionnaire. | | | | |
| Location | | Date | | |
| Study par | ticipant's signature | Responsible study physician | | |
| Texted name | | Texted name | | |